CLINICAL TRIAL: NCT03135132
Title: Metabolomics Identifies Increases in Acylcarnitine Profiles in Plasma of Overweight Subjects in Response to Mild Weight Loss
Brief Title: The Effect of Mild Weight Loss on Circulating Metabolite Profiles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Wt loss_metabolites
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Visceral Fat; Weight Loss
Keywords: High visceral fat; Low calorie diet; Mild weight loss; Metabolomics; Metabolites; Acylcarnitines
MeSH Terms: conditions — Weight Loss | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Usual dietary intake group
  Interventions: Behavioral: Control group
- LCD group (Experimental): Low calorie diet (LCD) group (300kcal/day intake reduction)
  Interventions: Behavioral: LCD group

INTERVENTIONS:
Behavioral: Control group — Recommend to consume usual diet during 12-week study period
  Arms: Control group
Behavioral: LCD group — Recommended to reduce calorie intake (a 300 kcal/day); educated to take out 1/3 of a bowl of rice from per meal a day for an easier application of 100kcal deficits, thereby reducing a 300kcal/3 meal/day
  Arms: LCD group

SUMMARY:
To determine whether low calorie diet (LCD)-induced weight reduction caused changes in plasma metabolites and metabolic traits from baseline.

DETAILED DESCRIPTION:
Over a 12-week clinical intervention period, a randomized, controlled study was carried out; overweight subjects consumed a LCD (approximately 300kcal/d deficit, n=47) or a weight-maintenance diet (control, n=50) were included for analyzing plasma samples and metabolites using an ultra-performance liquid chromatography and mass spectrometry (UPLC-LTQ/Orbitrap MS).

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* 20-65 years old
* Males and females
* Overweight (25.0 kg/m²≤ Body mass index <30 kg/m²)
* Nondiabetic (Fasting glucose <126 mg/dL)

Exclusion Criteria:

* Unstable body weight (body weight change >1 kg within 3 months before screening)
* Consumption of medication that affects body weight or energy expenditure
* Pregnancy or breast-feeding
* Hypertension, type 2 diabetes, cardiovascular disease, cerebrovascular disease, or thyroid disease
* Liver disease, kidney disease, or gastrointestinal disease
* Acute or chronic infections
* Any acute or chronic disease requiring treatment

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Visceral fat area at L4 (CT) | At baseline
Visceral fat area at L4 (CT) | At 12-week follow-up
Change in visceral fat area at L4 from baseline | At baseline and 12-week follow-up
Putatively identified plasma metabolites (Normalized peak intensities) | At baseline
Putatively identified plasma metabolites (Normalized peak intensities) | At 12-week follow-up
Changes in putatively identified plasma metabolites (Normalized peak intensities) from baseline | At baseline and 12-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, PhD, Principal Investigator — Yonsei University
Locations (1):
- Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jang HY, Han Y, Yoo HJ, Lee JH, Kim M. Effects of short-term dietary restriction on plasma metabolites and the subcutaneous fat area according to metabolic status in obese individuals: a case-control study. Diabetol Metab Syndr. 2021 Jun 7;13(1):62. doi: 10.1186/s13098-021-00679-8. PMID 34099056
- [Derived] Kang M, Yoo HJ, Kim M, Kim M, Lee JH. Metabolomics identifies increases in the acylcarnitine profiles in the plasma of overweight subjects in response to mild weight loss: a randomized, controlled design study. Lipids Health Dis. 2018 Oct 15;17(1):237. doi: 10.1186/s12944-018-0887-1. PMID 30322392